CLINICAL TRIAL: NCT02852044
Title: The Influence of Sampling Site When Assessing Glucose Tolerance or Insulin Sensitivity With Oral Glucose Ingestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Lecturer, University of Bath
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RE-CP
Record Dates: First submitted 2016-07-28; First posted 2016-08-02 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Hyperglycemia; Insulin Sensitivity
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance | interventions — RE1-silencing transcription factor; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rest (Active Comparator): Remain rested prior to the oral glucose tolerance test
  Interventions: Behavioral: Rest; Other: Dorsal Hand Vein Cannulation (heated hand technique); Other: Venous Cannulation
- Exercise (Experimental): Complete exercise prior to the oral glucose tolerance test
  Interventions: Behavioral: Exercise; Other: Dorsal Hand Vein Cannulation (heated hand technique); Other: Venous Cannulation

INTERVENTIONS:
Behavioral: Rest — Allowed to watch television or read for one hour prior to oral glucose tolerance test
  Arms: Rest
Behavioral: Exercise — One hour of cycling at 50% of maximal power output
  Arms: Exercise
Other: Dorsal Hand Vein Cannulation (heated hand technique)
Other: Venous Cannulation

SUMMARY:
For decades, it has been known that post-meal blood glucose concentrations were associated with the risk of T2D, which was reflected in early diagnostic guidelines. The oral glucose tolerance test (OGTT) has been used since at least 1923 and has remained the most common test for assessing glucose tolerance. Arterial blood (or arterialised blood using heated hand technique) is most appropriate for determining glucose tolerance and insulin sensitivity since this best represents the concentrations of metabolites and hormones that peripheral tissues are exposed to. It is essential to investigate whether venous blood (sometimes used during an OGTT) is representative of arterialised blood during an OGTT, and under different metabolic conditions.

The investigators want to understand whether OGTT-derived insulin sensitivity indices differ from venous and arterialised blood; and 2) investigate whether metabolic status (i.e. rest vs lower-limb exercise) influences the difference between forearm venous and arterialised concentrations of glucose and insulin during an OGTT.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-49 years
* Able and willing to safely comply with all study procedures
* Able to provide written informed consent for participation

Exclusion Criteria:

* Diagnosis of any bleeding disorder or taking medication which impacts blood coagulation
* The presence of any contraindications to maximal exercise testing, as determined using a physical activity readiness questionnaire (PAR-Q).
* Any diagnosis of metabolic disease (i.e. cardiovascular disease or type 2 diabetes).

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Postprandial plasma glucose concentrations (area under the concentration-time curve) | 120 mins
OGTT-derived insulin sensitivity | 120 mins

SECONDARY OUTCOMES:
Fasting plasma glucose concentrations | 5 mins
Fasting plasma insulin concentrations | 5 mins
Fasting plasma lactate concentrations | 5 mins
Fasting plasma triglyceride concentrations | 5 mins
Postprandial plasma lactate concentrations (area under the concentration-time curve) | 120 mins
Postprandial plasma triglyceride concentrations (area under the concentration-time curve) | 120 mins
Substrate utilization for energy provision | 180 mins
Postprandial plasma insulin concentrations (area under the concentration-time curve) | 120 mins

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nauck MA, Liess H, Siegel EG, Niedmann PD, Creutzfeldt W. Critical evaluation of the 'heated-hand-technique' for obtaining 'arterialized' venous blood: incomplete arterialization and alterations in glucagon responses. Clin Physiol. 1992 Sep;12(5):537-52. doi: 10.1111/j.1475-097x.1992.tb00357.x. PMID 1395446
- [Background] Liu D, Moberg E, Kollind M, Lins PE, Adamson U, Macdonald IA. Arterial, arterialized venous, venous and capillary blood glucose measurements in normal man during hyperinsulinaemic euglycaemia and hypoglycaemia. Diabetologia. 1992 Mar;35(3):287-90. doi: 10.1007/BF00400932. PMID 1563586